CLINICAL TRIAL: NCT00943332
Title: Pediatric Femur Research Project
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Missouri-Columbia (Other); Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Other Study IDs: 09-0819-201105030
Record Dates: First submitted 2009-07-17; First posted 2009-07-22 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Femur Fracture
Keywords: Orthopedic Procedures; Fracture Fixation, Internal; Fracture Fixation, External; femur fracture; pediatrics
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- spica casting
  Interventions: Procedure: femur fracture repair
- intramedullary nailing
  Interventions: Procedure: femur fracture repair
- submuscualr plating
  Interventions: Procedure: femur fracture repair

INTERVENTIONS:
Procedure: femur fracture repair — all participants will have undergone surgical intervention to repair a femur fracture, the investigators will simply be collecting data after the procedure; participants will not be consented until after the procedure

SUMMARY:
Current treatment protocol for pediatric femoral shaft fractures is immediate spica casting for patients 6 years and younger and for patients over 6 years and older is percutaneous or open placement of titanium elastic intramedullary nails. The investigators would like to evaluate the current treatment protocol by comparing those patients 6 years and younger treated with closed reduction and spica casting to those 6 years and younger treated with percutaneous pinned with titanium elastic intramedullary nails or submuscular plating. The investigators will be comparing their post-operative functional level, pain management, impact on family and complications through chart and x-ray reviews. The goal is to improve patient care pre and post-operatively for those who have sustained a femoral shaft fracture 6 years old and younger and increase the knowledge of those residents/physicians who care for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Child diagnosed with femur fracture between the ages of 2-6 years old
* Patient will undergo surgical intervention for a femur fracture (e.g., submuscular plating, Nancy nailing, casting )

Exclusion Criteria:

* Parent refusal to participate for any reason
* Children with neuromuscular disorders having a Gross Motor Function Classification greater than 3
* Pathologic fracture

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients will have undergone of the following interventions for the treatment of the femur fracture: spica casting, nancy nailing, or submuscular plating, by a participating physician in the trial. All of these treatments are considered standard of care for this pediatric population.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2009-06; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Impact on family | 6 months

SECONDARY OUTCOMES:
post-operative functional level | 1 year
pain management | 6 weeks
complications | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: J. Eric Gordon, MD, Principal Investigator — Washington Univeristy
Locations (3):
- United States (3):
  - Children's Hospital - University Missouri, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - St. Louis Childrens Hospital, St Louis, Missouri